CLINICAL TRIAL: NCT05931341
Title: The Effects of Oral Adminstration of Softgel Capsule Including Rosemary Extract on Pharmacokinetic Profile in Healthy Adults
Brief Title: Pharmacokinetic Profile of Rosemary Extract Supplement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CJ CheilJedang (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CJFNT000001
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — rosemary leaf extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dosage 1 (Experimental)
  Interventions: Dietary Supplement: Rosemary extract
- Dosage 2 (Experimental)
  Interventions: Dietary Supplement: Rosemary extract
- Dosage 3 (Experimental)
  Interventions: Dietary Supplement: Rosemary extract

INTERVENTIONS:
Dietary Supplement: Rosemary extract — Softgel capsule including rosemary extract

SUMMARY:
This study is a clinical trial to observe changes in biomarkers in the blood at pre- and post-supplementation of rosemary extract in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged between 25 and 55 years
* Non-smoker
* Body Mass Index (BMI) between 20 and 30 kg/m2

Exclusion Criteria:

* Any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, endocrine, metabolic, hematological, neurologic, psychiatric, systemic or infectious disease

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Concentration in plasma | 24 hours

IPD SHARING:
Plan to Share IPD: No